CLINICAL TRIAL: NCT04644926
Title: Effects of Remote Ischemic Conditioning on Microcirculatory Alterations in Patients With Sepsis
Brief Title: The Effect of Remote Ischemic Conditioning on the Microcirculation in Sepsis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Andrius Pranskunas, professor, Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE-2-78
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Septic Shock; Sepsis
Keywords: Microcirculation; Remote ischemic conditioning; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote ischemic conditioning (Experimental): Remote ischemic conditioning (RIC) is performed at inclusion and repeated 12 h and 24 h later.
  Interventions: Procedure: Remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) procedure comprise three repetitions of brachial cuff inflation to 200 mmHg for five minutes following deflation to 0 mmHg for another five minutes. The procedure overall took 30 minutes.

SUMMARY:
This study is an evaluation of the effect of Remote ischemic conditioning on sublingual microcirculation in patients with sepsis.

DETAILED DESCRIPTION:
This prospective open-label trial is performed in mixed ICU in a tertiary teaching hospital. Investigators include patients with sepsis or septic shock within the first 24 h after ICU admission. Remote ischemic conditioning (RIC) procedure comprise three repetitions of brachial cuff inflation to 200 mmHg for five minutes following deflation to 0 mmHg for another five minutes. The procedure overall took 30 minutes. RIC is performed at inclusion and repeated 12 h and 24 h later. Sublingual microcirculatory measurements are obtained before and after each RIC procedure, using incidence dark field (IDF) device.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis or septic shock within the first 24 h after ICU admission.

Exclusion Criteria:

* age < 18 years,
* pregnancy,
* advanced malignancy,
* peripheral artery disease affecting both arms,
* oral mucosal inflammation or injury or technical difficulties in obtaining sublingual images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Microvascular flow index (MFI) and Proportion of perfused small vessels (PPV) | 30 minutes
  The differences in MFI and PPV between pre- and post-RIC performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Lithuanian university of health sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiudulaite I, Belousoviene E, Vitkauskiene A, Pranskunas A. Effects of remote ischemic conditioning on microcirculatory alterations in patients with sepsis: a single-arm clinical trial. Ann Intensive Care. 2021 Apr 7;11(1):55. doi: 10.1186/s13613-021-00848-y. PMID 33829305